CLINICAL TRIAL: NCT04031092
Title: Use of Wearable Tech to Increase Physical Activity in Inpatient Rehabilitation for Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/800
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Chronic Pain; Musculoskeletal Pain
Keywords: Exercise; Biomedical Technology
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain; Motor Activity | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: A parallel group design with two groups
Who Masked: Investigator
Masking Description: The researchers performing the analyses will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wearable tech with feedback (Experimental): This group will be wearing an activity measurement device (wristband) and receive feedback about their activity level through a mobile application while taking part in a traditional inpatient rehabilitation program for patients with chronic pain.
  Interventions: Device: Wearable tech with feedback; Behavioral: Rehabilitation program
- Wearable tech without feedback (Active Comparator): This group will be wearing the same the activity measurement device as the intervention group, but they will not receive any feedback about their activity level. They will not have access to the mobile application. They will take part in the same rehabilitation program as the intervention group.
  Interventions: Device: Wearable tech without feedback; Behavioral: Rehabilitation program

INTERVENTIONS:
Device: Wearable tech with feedback — An armwrist device measuring physical activity level. The user will receive information about their physical activity level through their smartphone.
  Arms: Wearable tech with feedback
Device: Wearable tech without feedback — An armwrist device measuring physical activity level, no reporting back to the user.
  Arms: Wearable tech without feedback
Behavioral: Rehabilitation program — traditional inpatient rehabilitation program.

SUMMARY:
The aim of this project is to evaluate whether use of wearable tech increases levels of physical activity in patients participating in inpatient rehabilitation for chronic pain.

DETAILED DESCRIPTION:
Chronic pain is a vast problem with profound consequences for individuals and societies. Exercise and physical activity is an important part of the treatment for chronic pain. Use of wearable tech might be a way to help facilitate physical activity in patients with chronic pain. Here it will be evaluated whether use of wearable tech giving feedback about the user's activity level increases physical activity in patients participating in inpatient rehabilitation for chronic pain. The control group will be wearing the same wearable tech as the intervention group, but they will not receive any feedback about their activity level.

The feedback application will give participants in the intervention group information about the number of PAI they earn each week. PAI is short for personal activity Intelligence. You earn PAI points every time your heart rate increases: The higher heart rate, the faster you earn PAI. Previous research have shown that those who achieve 100 PAI or more every week over time live for an average of more than eight years longer than others.

During the study all participants will take part in a traditional inpatient rehabilitation program. The program consist of two periods at the rehabilitation center with two weeks at home in-between. The study will take place during the two periods at the senter and the period at home. Time spent on physical activity and number of earned PAI's will be counted during the period at home.

ELIGIBILITY:
Inclusion Criteria:

* taking part in inpatient rehabilitation at Unicare Helefort Rehabilitation center for chronic pain.

Exclusion Criteria:

* not having a smartphone (will not be able to access the mobile application).
* using a wheelchair (the technology will be not able to measure activity correctly)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Activity level | 2 weeks (time period at home between two stays at the rehabilitation center)
  Time spent in moderate to vigorous physical activity (minutes per day)
Number of PAIs | 2 weeks (time period at home between two stays at the rehabilitation center)
  mean number of Personal Activity Intelligence (PAI) points achieved per week
Percentage achieving 100 PAIs per week | 2 weeks (time period at home between two stays at the rehabilitation center)
  Personal Activity Intelligence (PAI)

SECONDARY OUTCOMES:
oxygen uptake | 6 weeks (from inclusion to end of rehabilitation program)
  submaximal oxygen uptake measured by the Åstrand bicycle test (described in Textbook of work physiology by Astrand from 1986)
Anxiety and depression symptoms | 6 weeks (from inclusion to end of rehabilitation program)
  HSCL-25 questionnaire
Average pain | 6 weeks (from inclusion to end of rehabilitation program)
  Visual Analogue Scale (VAS). VAS is a straight horizontal line where the ends are defined as the extreme limits from the left (0-no pain) to the right (100-worst imaginable pain). The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain.
Health related quality of life | 6 weeks (from inclusion to end of rehabilitation program)
  EQ5D questionnaire
Body weight | 6 weeks (from inclusion to end of rehabilitation program)
  body weight in kilograms
Body Mass Index score | 6 weeks (from inclusion to end of rehabilitation program)
  weight in kilograms divided by height in metres squared

CONTACTS AND LOCATIONS:
Overall Officials: Lene Aasdahl, PhD MD, Principal Investigator — National Taiwan Normal University; Jorunn Helbostad, Dr Philos, Study Director — Norwegian University of Science and Technology
Locations (1):
- Unicare Helsefort, Rissa, Norway

IPD SHARING:
Plan to Share IPD: No